CLINICAL TRIAL: NCT00778479
Title: Evaluation of the Safety of Sepraspray in Open Abdominal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by Sponsor: see details below
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSPRAY00508
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Adhesion Prevention (Abdominal)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sepraspray (Experimental): Receive Sepraspray
  Interventions: Device: Sepraspray
- Control (No Intervention): no treatment

INTERVENTIONS:
Device: Sepraspray — Max. 10g of Sepraspray
  Arms: Sepraspray

SUMMARY:
This study will examine the Performance of Sepraspray in Patients undergoing open abdominal surgery

NOTE regarding reason for study termination:

A patient death reported during the trial warranted temporary suspension for review by the independent data review committee. Although the committee recommended continuing enrollment, enrollment was electively terminated by the sponsor.

A preliminary analysis did not identify any new risk that was not listed on the investigational labeling for this product. A full analysis of the results is expected to allow characterization of the risk/benefit and clinical utility of the product in the exposed patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and over that require open abdominal surgery

Exclusion Criteria:

* Patients who are pregnant or have ongoing abdominal abscess or bacterial peritonitis or have infectious complications from a previous laparectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- France (4):
  - Chu Hotel Dieu, Clamond
  - CHRU de Lille, Hopital Huriez, Lille
  - Hopital de la Croix Rousse, Lyon
  - Hopital Lariboisiere, Paris
- Sweden (3):
  - University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala